CLINICAL TRIAL: NCT02036749
Title: Ultrasound-guided Quadratus Lumborum Block for Postoperative Pain Relief After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Krohg, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2013/1293
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- quadratus lumborum block (nerve block) (Active Comparator): quadratus lumborum block with ropivacaine
  Interventions: Procedure: nerve block
- sham block (Placebo Comparator): QL block with saline
  Interventions: Procedure: nerve block

INTERVENTIONS:
Procedure: nerve block — quadratus lumborum block
  Other Names: quadratus lumborum block

SUMMARY:
The Quadratus Lumborum (QL) Block is an ultrasound-guided technique described by Rafael Blanco in 2007. The nerves to the lower abdominal wall can be anesthetized by injecting local anesthetics close to the anterior border of the quadratus lumborum muscle. In our randomized, controlled, double-blinded study ultrasound-guided QL-blocks in 20 female patients after cesarean delivery will be compared with a placebo control group of 20 patients to investigate analgesic consumption, pain level, opioid related side effects and mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cesarean delivery
* American Society of Anesthesiologists classification (ASA) < 3
* adequate communication skills
* Body mass index < 32

Exclusion Criteria:

* ASA > 2
* chronic pain
* neurological illness/ neuropathy
* contraindication against local anesthetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 48 hours

SECONDARY OUTCOMES:
pain level (NRS) | 48 hours

OTHER OUTCOMES:
time to mobilization | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anders Krohg, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway